CLINICAL TRIAL: NCT06971887
Title: Embedding Health Literacy Best Practices: A Feasibility Study Using the Clear Communication of Laboratory Test Results (CCLR) Template
Brief Title: Feasibility Study of Use and Acceptability of New Clear Communication of Lab Test Results (CCLR) Letter for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Nancy Morris, Professor, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 00000965
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Communication
Keywords: Health Literacy; Lab test results communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: First 30 participants received standard of care; 2nd 30 participants received the Clear Communication of Laboratory Result templated result note
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants received the standard communication letter for result of blood test (No Intervention): Providers send their usual result note related to a blood test
- Clear Communication of Lab Test Result letter (Experimental): Participants received the results of their blood test on the Clear Communication of Lab Test Results (CCLR) letter
  Interventions: Other: Clear Communication of Lab Test Result letter

INTERVENTIONS:
Other: Clear Communication of Lab Test Result letter — The Clear Communication of Lab Test Result letter (CCLR) was designed using clear communication and health literacy best practices to explain test done, meaning of results, and any future action recommended.
  Arms: Clear Communication of Lab Test Result letter

SUMMARY:
This study will try out a new way of writing a blood test result letter to patients explaining the results in a way to help them understand what the results mean and any next steps to be taken.

DETAILED DESCRIPTION:
The primary goal of this study was to help healthcare providers more effectively communicate the meaning of laboratory test results and any need for follow-up, facilitating patient engagement in their healthcare. The investigators propose that using an innovative laboratory test result template integrating health literacy best practices, specifically the Clear Communication of Lab Results (CCLR) template, has the potential to improve health outcomes and health care processes. The purpose of this study was to create and assess the feasibility of using the CCLR template for 3 common laboratory tests to increase knowledge and confidence, decrease anxiety, activate follow-up, and improve satisfaction among older adults.

ELIGIBILITY:
Inclusion Criteria:

* age 70 or older
* English fluency
* order for CBC, BMP, or FLP
* capacity to provide informed consent
* willingness to participate in follow-up phone survey

Exclusion Criteria:

* provider determined potential participant does not have cognitive capacity to read or understand communication about lab test results

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Recruitment | 18 months
  Investigators will recruit participants for the study and providers will use the Clear Communication of Lab Test Result Letter

SECONDARY OUTCOMES:
Global Anxiety-Visual Scale | 2 weeks after blood test was drawn
  Measure of anxiety after receiving the lab result letter. The minimum value is zero (0) and the maximum value is 100; higher scores mean greater anxiety.
Confidence | 2 weeks after blood test was drawn
  Visual analogue scale to assess confidence in understanding meaning of lab test result. The minimum score is 1 (not at all satisfied) and the maximum score is 10 (extremely satisfied). Higher score reflects higher confidence.
Comprehension of follow-up plans | 2 weeks after blood test was drawn
  Yes/No response to question, Was it clear if there were any next steps participant needs to do related to the blood test results?
Patient Satisfaction | 2 weeks after blood test was drawn
  Visual analogue scale response to question, how satisfied was the participant with the letter describing lab test results? Minium response is one (1) not at all satisfied and the maximum response is 10, extremely satisfied. A higher score reflects higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Morris, PhD, RN, ANP-BC, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This was a feasibility trial and undertaken to learn what should be changed for a larger, powered study.